CLINICAL TRIAL: NCT05214703
Title: The Effect of Cold Therapy on Pain and Anxiety During the Implanted Port Catheter Removal Procedure
Brief Title: The Effect of Cold Therapy on Pain and Anxiety During the Implanted Port Catheter Removal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yuksek Ihtisas University (Other)
Responsible Party: Principal Investigator, Arzu Bahar, assistant professor, Yuksek Ihtisas University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: YuksekIU-ABAHAR-002
Record Dates: First submitted 2022-01-14; First posted 2022-01-31 (Actual); Last update posted 2022-01-31 (Actual); Status verified 2022-01

CONDITIONS: Pain; Anxiety
Keywords: Cancer; Venous Port Catheter; Cold Therapy; Pain; Anxiety
MeSH Terms: conditions — Pain; Anxiety Disorders; Neoplasms

STUDY DESIGN:
Intervention Model Description: Parallel Assignment a clinical trial with experimental and control groups with
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- cold therapy (Experimental): Pain scores were measured with a visual analog scale (VAS) before the port catheter was removed from the patients in the experimental group. Before the port catheters were removed, cold application with an ice pack was applied to the patients whose first visual analog scale measurement was made by the researchers. The cold application was terminated an average of 15 minutes after the body temperature decreased by 1 °C.
  Interventions: Other: cold therapy application
- no intervention (No Intervention): The patients in the control group did not receive any intervention before and after port catheter removal.

INTERVENTIONS:
Other: cold therapy application — cold therapy
  Arms: cold therapy

SUMMARY:
This study was conducted as a quasi-experimental study to examine the effect of cold therapy on pain and anxiety during venous port catheter removal.

DETAILED DESCRIPTION:
Pain and anxiety experienced during diagnosis and treatment in cancer patients affect the physical, psychological, and interpersonal well-being of individuals and affect their lives in all aspects. Nurses play a very important role in pain control. Pain control is very important in terms of ensuring the comfort of patients and increasing their quality of life. In order to provide this control; nurses can use non-pharmacological treatment methods that they can apply independently in pain management. Patients experience procedural pain during insertion and removal of an implantable port catheter, which is one of the painful invasive procedures that are placed under the skin with a small incision, and insertion of a needle into the port catheter. When the literature is examined, it is seen that there are a limited number of studies in which non-pharmacological methods are used in the control of pain and anxiety related to the implantable venous port catheter procedure, and in these studies, distraction, music therapy, and inhaler aromatherapy. However, no study was found in which cold application was used to reduce the pain and anxiety caused by the removal of the port catheter in cancer patients. Therefore, the aim of the study is to evaluate the effectiveness of cold application on procedural pain and anxiety associated with port catheter removal, which is frequently used in the treatment of cancer patients. Cold therapy as an independent nursing intervention in reducing anxiety and pain management during port catheter removal in cancer/oncology patients; can be transferred to clinical practice by oncology nurses, improving the quality of nursing care, ensuring patient safety, and increasing patient satisfaction. In addition, the results of the research may contribute to the literature in terms of increasing evidence-based information on the use of the cold application in procedural pain and anxiety control in cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of cancer disease
* 18 years and over
* no analgesic medication before three hours before the catheter removal procedure
* conscious and cooperative
* no communication problems
* no visual no vision problems
* with stable vital signs
* without a diagnosis of anxiety disorder
* volunteer participation

Exclusion Criteria:

* Body mass index less than 18.5
* receiving Oxaliplatin infusions before venous port catheter removal

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 112 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2018-09-01 (Actual)

PRIMARY OUTCOMES:
Vertical Visual Analog Scale(VAS) | 20 minutes
  Pain scores of the experimental and control groups were evaluated with VAS. The pain scores in both groups were shown to the patients by the researchers by showing the VAS, and they were asked to show at which point they experienced pain. The VAS scores of the patients in both groups were measured 10 minutes before the port catheter was removed (1st measurement), immediately after the catheter was removed (2nd measurement), and 10 minutes after the catheter was removed (3rd measurement).
  Pain intensity was measured by using a vertical visual analog scale(VAS) from "0 to 10", with high numbers meaning greater pain intensity. Iıt is indicated that compared with other tools, the vas is more sensitive and reliable in the measurement of pain intensity. Pain intensity can be categorized as mild (score, 1-3), moderate (score, 4-6), and severe (score, 7-10) according to the scale.

SECONDARY OUTCOMES:
The StateTrait Anxiety Inventory(STAI-I) | 20 minutes
  The scores of the State-Trait Anxiety Inventory(STAI-I) Anxiety levels of the experimental and control groups were evaluated with STAI-I. The STAI-I scores of patients in both groups were measured 10 minutes before port catheter removal (1st measurement), and 10 minutes after catheter removal (2nd measurement).
  The patient's level of anxiety was evaluated by the State-Trait Anxiety Inventory(STAI-I.). While the first 20 items in the scale determine the state anxiety level, the second 20 items evaluate the trait anxiety level. The scores obtained from both scales theoretically vary between 20-80. In terms of anxiety levels in STAI-I, "0-19 points" from the scale, no anxiety, "20-39" points mild, "40-59" points moderate, "60-79" points severe, "80" score is evaluated as the level of panic and severe anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Arzu bahar, PhD, Principal Investigator — Yuksek Ihtisas University
Locations (1):
- Arzu Bahar, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bahar A, Aktas D, Sonmez M. Effects of Cold Therapy on Pain and Anxiety During Needle Removal From Implanted Ports. J Infus Nurs. 2023 Jan-Feb 01;46(1):36-42. doi: 10.1097/NAN.0000000000000495. PMID 36571826